CLINICAL TRIAL: NCT04623034
Title: A Phase 1, Two Stage, Open Label, Randomized, Single Dose, Comparative Study to Evaluate the Safety and Pharmacokinetics of MSI-195 to a Commercial S-Adenosylmethionine Product in Healthy Volunteers
Brief Title: Evaluation of the Safety and Pharmacokinetics of MSI-195 to a Commercial S-Adenosylmethionine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MSI Methylation Sciences, Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MSI-CP.001.02
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Major Depressive Disorder
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: Stage 1 - single ascending dose, Stage 2 - crossover and food effect study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 400 mg MSI-195 - SAD (Experimental): 400 mg MSI-195 (within Stage 1, single ascending dose)
  Interventions: Drug: Ademetionine
- 800 mg MSI-195 - SAD (Experimental): 800 mg MSI-195 (within Stage 1, single ascending dose)
  Interventions: Drug: Ademetionine
- 1600 mg MSI-195 -SAD (Experimental): 1600 mg MSI-195 (within Stage 1, single ascending dose)
  Interventions: Drug: Ademetionine
- 800 mg MSI-195 - fasted (Experimental): 800 mg MSI-195 fed (within Stage 2, cross-over comparison)
  Interventions: Drug: Ademetionine
- 1600 mg SAM-e Complete TM - fasted (Experimental): 1600 mg SAM-e Complete (within Stage 2, cross-over comparison)
  Interventions: Drug: Ademetionine
- 800 mg MSI-195 - fed (Experimental): 800 mg MSI-195- fed (within Stage 2, fed arm)
  Interventions: Drug: Ademetionine

INTERVENTIONS:
Drug: Ademetionine

SUMMARY:
This study was a pharmacokinetic and safety evaluation of the S-adenosylmethionine formulation MSI-195, and a commercial comparator. The study was broken into two stages. The first stage was an exploratory single ascending dose design of MSI-195 in 8 healthy normal male volunteers. The second stage was a single dose evaluation, targeting 26 male and female volunteers at set doses of MSI-195 and commercial comparator in a cross-over design followed by a food effect study on MSI-195. Plasma samples were collected and assayed for S-adenosylmethionine. Pharmacokinetic parameters were calculated using that data.

DETAILED DESCRIPTION:
The study was focussed on the safety and pharmacokinetic evaluation of MSI-195; a novel patented formulation of S-adenosylmethionine. MSI-195 is a 400 mg dosage strength, tablet formulation comprising a core tablet, a seal coat and an enteric coat. The commercial comparator is SAM-e CompleteTM, manufactured by Pharmavite under the NatureMadeTM brand.

This study consisting of two stages. The first stage was an exploratory single ascending dose design of MSI-195 in 8 healthy normal male volunteers. The second stage was a more comprehensive single dose evaluation, targeting 26 male and female volunteers at set doses of MSI-195 and commercial comparator in a cross-over design followed by a food effect study on MSI-195.

Stage 1 design In each period of this stage of the study, ascending single doses of 400 mg, 800 mg and 1600 mg of MSI-195 was orally administered under fasted conditions, followed by 24 hours of blood draws at periodic intervals for the determination of plasma concentration of S-adenosylmethionine in a repeated-measure design. The drug administrations were separated by a wash-out of 7 calendar days.

Stage 2 design In the first 2 periods of this stage of the study, a single 800 mg dose of MSI-195 and a single 1600 mg dose of commercial comparator were orally administered under fasted conditions, in a 2-way crossover design. During the 3rd period, a single 800 mg dose of MSI-195 was administered under fed conditions to all subjects. The drug administrations were separated by a wash-out of 7 calendar days. For each dosing, subjects had periodic blood draws over a 24 hour period to determine the plasma concentration of S-adenosylmethionine as a function of time.

Male and female volunteers were included in the study. Subjects were in good health as determined by a medical history, complete physical examination (including vital signs), electrocardiogram (ECG), neurological examination and a panel of clinical laboratory tests.

Blood samples were collected and stored frozen until assayed. The samples were assayed for S-adenosylmethionine using a validated HPLC method with MS/MS detection.

For pharmacokinetic assessments, the main absorption and disposition parameters were calculated using a non-compartmental approach with a log-linear terminal phase assumption. The pharmacokinetic parameters of this trial were Cmax, Tmax, AUCT, AUC∞, AUCT/∞, Kel and T½el.

The safety parameters assessed included the occurrence of adverse events, the measurement of clinical laboratory parameters, vital signs, neurological function tests, physical examination and ECG

ELIGIBILITY:
Inclusion Criteria:

* Volunteers meeting all of the following criteria will be considered for enrollment in the study:

  1. Availability for the entire study period
  2. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
  3. Male or female volunteer (Male only for Stage 1 - Cohort 1)
  4. A female volunteer must meet one of the following criteria:

     1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens throughout her entire participation in the study. An acceptable method of contraception includes one of the following:

        * Abstinence from heterosexual intercourse
        * Systemic contraceptives (birth control pills, injectable/implantable /insertable hormonal birth control products, transdermal patch)
        * Intrauterine device
        * Condom with spermicide or
     2. Participant is of non-childbearing potential, defined as a female who had had a hysterectomy or tubal ligation, is clinically considered infertile or is in a menopausal state (at least 1 year without menses)
  5. Volunteer aged of at least 21 years but not older than 55 years
  6. Volunteer with a body mass index (BMI) greater than or equal to 18.50 and below 30.00 kg/m2
  7. Non- or ex smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 6 months before day 1 of this study.
  8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
  9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, ECG and urines)
  10. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer

The informed consent form must be signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

* Volunteers presenting any of the following will not be included in the study:

  1. Females who are pregnant or are lactating
  2. History of significant hypersensitivity to S-Adenosylmethionine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
  3. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
  4. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
  5. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
  6. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
  7. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec, QTc > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
  8. Presence or history of bipolar disorder
  9. Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
  10. Any clinically significant illness in the previous 28 days before day 1 of this study
  11. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
  12. Any history of tuberculosis and/or prophylaxis for tuberculosis
  13. Positive urine screening of alcohol and/or drugs of abuse
  14. Positive results to HIV Ag/Ac Combo, HBsAg (B) (hepatitis B) or anti-HCV (C) tests
  15. Females who are pregnant according to a positive serum pregnancy test
  16. Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
  17. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

No subjects will be allowed to enroll in this study more than once (i.e. if the study is conducted with more than 1 group).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04-17 (Actual); Primary Completion 2013-06-08 (Actual); Study Completion 2013-06-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-related adverse events (safety and tolerability) as measured by vital signs, ECG, laboratory tests, neurological function tests, and the occurance of adverse events | for 24 hours after dosing
  Incidence and severity of treatment-related adverse events determined by changes from screening (baseline) of findings from physical examination, vital signs, ECG, laboratory tests, neurological function tests, and the occurance of adverse events.
Pharmacokinetics was evaluated by measuring the systemic plasma concentration of ademetionine | for 24 hours after dosing
  plasma concentrations of ademetionine were measured as a function of time using a validated bioanalytical assay

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cameron BR, Ferreira L, MacDonald ID. Pharmacokinetic study of a novel oral formulation of S-adenosylmethionine (MSI-195) in healthy subjects: dose escalation, food effect and comparison to a commercial nutritional supplement product. BMC Pharmacol Toxicol. 2020 Dec 14;21(1):88. doi: 10.1186/s40360-020-00466-7. PMID 33317621